CLINICAL TRIAL: NCT04683809
Title: The Effect of Telerehabilitation on Quality of Life, Anxiety and Depression Levels in Children With Cystic Fibrosis and Their Caregivers
Brief Title: Effects of a Telerehabilitation Approach in Children With Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1442
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Cystic Fibrosis
Keywords: anxiety; depression; cystic fibrosis; caregiver; telerehabilitation
MeSH Terms: conditions — Cystic Fibrosis; Anxiety Disorders; Depression | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients in this group will attend telerehabilitation sessions.
  Interventions: Other: Telerehabilitation
- Control group (No Intervention): Patients in this arm will be subject to routine follow up.

INTERVENTIONS:
Other: Telerehabilitation — Patients will attend rehabilitation sessions through online programmes for rehabilitation
  Arms: Exercise group

SUMMARY:
Patients with cystic fibrosis aged 6-13 will be recruited and randomized into two groups: one will receive telerehabilitation sessions including postural, breathing and high-intensity interval training exercises and one will be subject to routine follow up. Exercise program will be applied three days a week for three months. Children will be assessed by pulmonary function tests, cystic fibrosis quality of life questionnaire, six minute walking test and anxiety and depression scale in children, while caregivers will be assessed by Beck depression scale and situational anxiety inventory.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed cystic fibrosis

Exclusion Criteria:

* Current pulmonary exacerbation
* Musculoskeletal problems hinder exercising
* No internet access
* Patients and parents do not consent to intervention

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cystic fibrosis quality of life questtionaire | 3 months
  Cystic fibrosis quality of life questtionaire

IPD SHARING:
Plan to Share IPD: Undecided